CLINICAL TRIAL: NCT00939809
Title: A Phase II Evaluation of a Urokinase-Derived Peptide (A6) in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: A6 in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0170N; NCI-2011-01927 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0170N; CDR0000644399; GOG-0170N (Other: Gynecologic Oncology Group); GOG-0170N (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2015-02

CONDITIONS: Fallopian Tube Carcinoma; Malignant Ovarian Mixed Epithelial Tumor; Ovarian Brenner Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Primary Peritoneal Carcinoma; Recurrent Ovarian Carcinoma; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Brenner Tumor; Ovarian Neoplasms

ARMS (1):
- Treatment (urokinase-derived peptide A6) (Experimental): Patients receive A6 subcutaneously once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Urokinase-Derived Peptide A6; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Urokinase-Derived Peptide A6 — Given SC
  Other Names: A6; uPA-derived Peptide A6
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well A6 works in treating patients with persistent or recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer. A6 may stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of A6, as measured by the 6-month progression-free survival (PFS) rate and objective tumor response (complete or partial) rate, in patients with persistent or recurrent ovarian epithelial, fallopian tube, or primary peritoneal carcinoma.

II. To determine the frequency and severity of adverse events as assessed by CTCAE v3.0.

SECONDARY OBJECTIVES:

I. To characterize the duration of PFS and overall survival. II. To identify biomarkers of drug effect on peripheral blood mononuclear cells (PBMCs).

TERTIARY OBJECTIVES:

I. To explore whether genes identified as being up- or down-regulated by exposure of human PBMCs to A6 in vitro are also up- or down-regulated following treatment of patients with A6 in vivo.

II. To explore whether there is an association between the expression of candidate A6 receptors in the tumor prior to treatment with A6 (as determined by IHC) and response and PFS.

III. To explore whether there is an association between change in expression of candidate biomarkers in PBMCs between 0-24 hours following the first dose of A6 and response and PFS.

IV. To explore whether there is an association between change in expression of candidate biomarkers in PBMCs over the course of the first one month cycle (course 1) and response and PFS.

V. To determine whether there is an association between plasma A6 levels measured on days 2 (24 hours after the first dose and 4 hours after the second dose) and 8 (prior to injection of A6) of course 1 and levels of expression of candidate biomarkers in PBMCs collected on the same days.

VI. To explore whether there is an association between plasma A6 levels measured on days 2 (24 hours after the first dose and 4 hours after the second dose) and 8 (prior to injection of A6) of course 1 and response and PFS.

VII. To explore whether there is an association between candidate serum biomarkers and response and PFS over the course of A6 treatment.

OUTLINE: This is a multicenter study.

Patients receive A6 subcutaneously once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed persistent or recurrent ovarian epithelial, fallopian tube, or primary peritoneal carcinoma, including any of the following epithelial cell types:

  * Serous adenocarcinoma
  * Endometrioid adenocarcinoma
  * Mucinous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Transitional cell carcinoma
  * Malignant Brenner tumor
  * Adenocarcinoma not otherwise specified
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must have ≥ 1 target lesion to assess response as defined by RECIST criteria

  * Tumors within a previously irradiated field are designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence of disease ≥ 90 days following completion of radiotherapy
* Must not be eligible for a higher priority GOG clinical trial, if one exists (i.e., any active GOG Phase III clinical trial for the same patient population)
* Must have received 1 prior platinum-based chemotherapeutic regimen containing carboplatin, cisplatin, or another organoplatinum compound for management of primary disease

  * Initial treatment may have included high-dose therapy, consolidation therapy, non-cytotoxic therapy, or extended therapy administered after surgical or non-surgical assessment
  * One additional cytotoxic regimen for management of recurrent or persistent disease allowed
  * Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease) must have a platinum-free interval of < 12 months, have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* GOG performance status 0-2 (for patients who received 1 prior regimen) OR 0-1 (for patients who received 2 prior regimens)
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able and willing to self-administer daily subcutaneous (SC) injections or has a caregiver who is willing and able to administer daily SC injections
* No active infection requiring antibiotics, except uncomplicated urinary tract infection
* No neuropathy (sensory and motor) > grade 2, according to CTCAE v3.0
* No other invasive malignancies within the past 5 years, except for non-melanoma skin cancer
* No history of sensitivity to A6
* No active gastrointestinal bleeding within the past month
* No other disease that, in the opinion of the investigator, could jeopardize patient safety or interfere with study objectives
* No concurrent amifostine or other protective reagents
* Recovered from prior surgery, radiotherapy, or chemotherapy
* No prior non-cytotoxic therapy for management of recurrent or persistent disease

  * Prior biologic (non-cytotoxic) therapy as part of primary treatment regimen allowed
* At least 1 week since prior hormonal therapy directed at the malignant tumor
* At least 3 weeks since any other prior therapy directed at the malignant tumor, including immunological agents
* More than 2 weeks since prior major surgical procedure
* More than 5 years since prior radiotherapy to any portion of the abdominal cavity or pelvis other than for the treatment of ovarian, fallopian tube, or primary peritoneal cancer
* More than 3 years since prior radiotherapy for localized cancer of the breast, head and neck, or skin AND remains free of recurrent or metastatic disease

  * Patients with ductal breast carcinoma in situ may have undergone localized radiotherapy within the past 3 years
* More than 5 years since prior chemotherapy for any abdominal or pelvic tumor other than for the treatment of ovarian, fallopian tube, or primary peritoneal cancer
* More than 3 years since prior adjuvant chemotherapy for localized breast cancer AND remains free of recurrent or metastatic disease
* More than 30 days since prior investigational drugs
* No prior A6
* No prior radiotherapy to > 25% of marrow-bearing areas
* No prior cancer treatment that would contraindicate study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, Principal Investigator — Gynecologic Oncology Group
Locations (16):
- United States (16):
  - Georgia Regents University Medical Center, Augusta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Stony Brook University Medical Center, Stony Brook, New York
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 7/6/2009 and closed to accrual on 1/4/2010.
Groups:
- A6 (Subcutaneous): 300 mg A6 Subcutaneously daily (2 injections of 150 mg) (cycle = 28 days) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | A6 (Subcutaneous)
Started | 31
Completed | 28 (Patients treated until disease progression; completed defined as off treatment due to progression.)
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | A6 (Subcutaneous)
Number analyzed (Participants) | 31
Age, Customized [Number; unit: participants]
  40-49 years | 1
  50-59 years | 11
  60-69 years | 17
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since study entry, or unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
  CT scan or MRI is used to follow lesion for measurable disease every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels. Responses must be confirmed by repeat imaging 4 weeks following documentation of response.
Time Frame: Scans to assess progression were done every other cycle for the first 6 months.
Population: Eligible and treated participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | A6 (Subcutaneous)
Number analyzed (Participants) | 31
percentage of participants | 6.5 [1.2 to 18.9]

2. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Per RECIST v1.0 for target lesions and assessed by MRI or CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  CT scan or MRI is used to follow lesion for measurable disease every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels. Responses must be confirmed by repeat imaging 4 weeks following documentation of response.
Time Frame: Scans to assess response were done every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels.
Population: Eligible and treated participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | A6 (Subcutaneous)
Number analyzed (Participants) | 31
percentage of participants | 0 [0 to 9.2]

3. Primary Outcome: Incidence of Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Time Frame: Every cycle during treatment (average collection time = 4 months)
Population: Eligible and Treated Patients
Measure: Count of Participants; unit: Participants
Arm/Group | A6 (Subcutaneous)
Number analyzed (Participants) | 31
Participants
  Constitutional | 2
  Gastrointestinal | 1
  Hemorrhage | 1

4. Secondary Outcome: Progression-free Survival
Description: as for outcome 1
Time Frame: as for outcome 2
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A6 (Subcutaneous)
Number analyzed (Participants) | 31
months | 2.0 [1.8 to 3.0]

5. Secondary Outcome: Overall Survival
Time Frame: Every other cycle, up to 5 years
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A6 (Subcutaneous)
Number analyzed (Participants) | 31
months | 10.6 [8.4 to NA] — NA (not applicable): insufficient number of participants with events.

6. Secondary Outcome: Biomarkers of Drug Effect on Peripheral Blood Mononuclear Cells (PBMCs)
Description: Note: due to the limited activity of this agent, it was decided not to expend resources assaying the PBMCs. Data was not collected.
Time Frame: Day 1 prior to dosing; Day 2 prior to dosing and 4-hour post dosing; Day 8 prior to dosing.
Population: due to the limited activity of this agent, it was decided not to expend resources assaying the PBMCs.
Arm/Group | A6 (Subcutaneous)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were queried for and collected every cycle for the duration of treatment.
Arm/Group | A6 (Subcutaneous)
Serious Adverse Events (participants affected / at risk) | 9/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A6 (Subcutaneous) (N=31)
Death No Ctcae Term - Sudden Death (General disorders) | 1
Distention (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 2
Hemorrhage, Cns (Vascular disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Nerve-Peripheral (Infections and infestations) | 1
Pain: Back (General disorders) | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A6 (Subcutaneous) (N=31)
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 5
Platelets (Blood and lymphatic system disorders) | 5
Leukocytes (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 17
Hypertension (Cardiac disorders) | 4
Sweating (General disorders) | 1
Weight Gain (General disorders) | 2
Fever (General disorders) | 1
Fatigue (General disorders) | 14
Insomnia (General disorders) | 2
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 3
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 2
Bruising (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Anorexia (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 1
Edema: Limb (Blood and lymphatic system disorders) | 2
Ast (Metabolism and nutrition disorders) | 2
Gfr (Metabolism and nutrition disorders) | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Alt (Metabolism and nutrition disorders) | 1
Alkaline Phosphatase (Metabolism and nutrition disorders) | 2
Bilirubin (Metabolism and nutrition disorders) | 1
Lipase (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1
Amylase (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 1
Mood Alteration - Anxiety (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 6
Flashing Lights/Floaters (Eye disorders) | 1
Pain - Other (General disorders) | 2
Pain: Pelvis (General disorders) | 1
Pain: Head/Headache (General disorders) | 3
Pain: Extremity-Limb (General disorders) | 1
Pain: Back (General disorders) | 6
Pain: Joint (General disorders) | 4
Pain: Bladder (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 13
Pain: Skin (General disorders) | 1
Pain: Muscle (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Leak, Gu - Urethra (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Bladder Spasm (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Note: due to the limited activity of this agent, it was decided not to expend resources assaying the PBMCs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No